CLINICAL TRIAL: NCT00098475
Title: A Randomized Phase III Study of CC-5013 Plus Dexamethasone Versus CC-5013 Plus Low Dose Dexamethasone in Multiple Myeloma With Thalidomide Plus Dexamethasone Salvage Therapy for Non-Responders
Brief Title: Lenalidomide and Dexamethasone With or Without Thalidomide in Treating Patients With Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-03150; NCI-2012-03150 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E4A03; CDR0000404161; E4A03 (Other: ECOG-ACRIN Cancer Research Group); E4A03 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: DS Stage I Multiple Myeloma; DS Stage II Multiple Myeloma; DS Stage III Multiple Myeloma
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; Thalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (lenalidomide, dexamethasone) (Active Comparator): Patients receive lenalidomide PO QD on days 1-21 and standard-dose dexamethasone PO QD on days 1-4, 9-12, and 17-20.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide
- Arm II (lenalidomide, low-dose dexamethasone) (Experimental): Patients receive lenalidomide and acetylsalicylic acid as in Arm I and low-dose dexamethasone PO QD on days 1, 8, 15, and 22.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide
- Arm III (thalidomide, dexamethasone) (Active Comparator): Patients with no response after treatment on Arm I: Patients receive thalidomide PO QD on days 1-28 and standard-dose dexamethasone PO QD on days 1-4, 9-12, and 17-20
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Thalidomide
- Arm IV (thalidomide, low-dose dexamethasone) (Experimental): Patients with no response after treatment on Arm II: Patients receive thalidomide as in arm III and low-dose dexamethasone PO QD on days 1, 8, 15, and 22.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Thalidomide

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Other: Laboratory Biomarker Analysis — Optional correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm I (lenalidomide, dexamethasone); Arm II (lenalidomide, low-dose dexamethasone)
Drug: Thalidomide — Given PO
  Other Names: (+)-Thalidomide; (-)-Thalidomide; .alpha.-Phthalimidoglutarimide; 2, 6-Dioxo-3-phthalimidopiperidine; Alpha-Phthalimidoglutarimide; Contergan; Distaval; Kevadon; N-(2,6-Dioxo-3-piperidyl)phthalimide; N-Phthaloylglutamimide; N-Phthalylglutamic Acid Imide; Neurosedyn; Pantosediv; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (+)-; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (-)-; Sedalis; Sedoval K-17; Sedoval K17; Softenon; Synovir; Talimol; Thalomid
  Arms: Arm III (thalidomide, dexamethasone); Arm IV (thalidomide, low-dose dexamethasone)

SUMMARY:
This randomized phase III trial studies lenalidomide and low-dose dexamethasone to see how well it works compared to lenalidomide and standard-dose dexamethasone, given with or without thalidomide, in treating patients with multiple myeloma. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Lenalidomide and thalidomide may also stop the growth of multiple myeloma by blocking blood flow to the cancer. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide, thalidomide, and dexamethasone together may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the response rate and toxicity of lenalidomide (CC-5013) plus dexamethasone (standard dose) versus CC-5013 plus low dose dexamethasone in patients with newly diagnosed myeloma at any time in the first 4 cycles of treatment and to determine if CC-5013 plus low dose dexamethasone will have similar response rate with lower toxicity (First Phase).

SECONDARY OBJECTIVES:

I. To evaluate the response rate of thalidomide plus dexamethasone (Thal/Dex) in patients with newly diagnosed myeloma who do not achieve a complete or partial response at any time in the first 4 cycles with the CC-5013 and dexamethasone combination in either of the two arms (First Phase).

II. To study the effect of CC-5013 on bone marrow microvessel density and angiogenesis grade, on plasma cell labeling index (PCLI), and on the expression of vascular endothelial growth factor (VEGF) and basic fibroblast growth factor (bFGF) in the marrow (First Phase).

III. To study the effect of CC-5013 and dexamethasone on bone marrow mesenchymal progenitor cells (MPCs) (First Phase).

IV. To evaluate in a separate expansion phase the efficacy of aspirin (325 mg/day) versus Coumadin (dose adjusted to maintain a target international normalized ratio [INR] of 2-3) in preventing deep vein thrombosis (DVT) in patients with newly diagnosed myeloma receiving CC-5013 plus standard dose dexamethasone.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21, and standard-dose dexamethasone PO QD on days 1-4, 9-12, and 17-20.

Arm II: Patients receive lenalidomide as in Arm I and low-dose dexamethasone PO QD on days 1, 8, 15, and 22.

In both arms, cycles repeat every 28 days in the absence of unacceptable toxicity or disease progression. Patients not responding at any point during the first 4 cycles of lenalidomide and dexamethasone are assigned to 1 of 2 salvage therapy arms. Patients who progress during treatment on Arms I or II have the option to register on salvage therapy Arms III or IV respectively.

Arm III (patients with no response after treatment on Arm I): Patients receive thalidomide PO QD on days 1-28 and standard-dose dexamethasone PO QD on days 1-4, 9-12, and 17-20.

Arm IV (patients with no response after treatment on Arm II): Patients receive thalidomide as in Arm III and low-dose dexamethasone PO QD on days 1, 8, 15, and 22.

In both salvage therapy arms, cycles repeat every 28 days in the absence of unacceptable toxicity or disease progression. After completion of 4 cycles of therapy, patients may undergo stem cell harvest (using growth factors only) for cryopreservation.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with symptomatic multiple myeloma within the past 90 days confirmed by the following:

  * Bone marrow plasmacytosis with >= 10% plasma cells or sheets of plasma cells or biopsy proven plasmacytoma which must be obtained within 4 weeks prior to randomization
  * Measurable levels of monoclonal protein (M protein): >= 1.0 g/dL on serum protein electrophoresis or >= 200 mg of monoclonal light chain on a 24 hour urine protein electrophoresis which must be obtained within 4 weeks prior to randomization; both serum protein electrophoresis (SPEP) and urine protein electrophoresis (UPEP) are required to be performed within 28 days prior to randomization; please note that if both serum and urine m-components are present, both must be followed in order to evaluate response
* Hemoglobin > 7 g/dL
* Platelet count > 75,000 cells/mm^3
* Absolute neutrophil count > 1000 cells/mm^3
* Creatinine < 2.5 mg/dL and creatinine clearance (measured or calculated) >= 60 mL/min
* Bilirubin =< 1.5 mg/dL
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) and serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 times the upper limit of normal
* Prior palliative and/or localized radiation therapy is permitted provided at least 4 weeks have passed from date of last radiation therapy to date of registration; patients with prior solitary plasmacytoma treated with radiation therapy with curative intent are eligible if the disease has now progressed to active multiple myeloma meeting all the eligibility criteria for this protocol
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days and again within 24 hours prior to starting cycle 1 of lenalidomide; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method (intrauterine device [IUD], birth control pills, tubal ligation or partner's vasectomy) and one additional effective method (condom, diaphragm or cervical cap); FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy starting 4 weeks prior to and while taking CC5013 or thalidomide and for four weeks after discontinuing this therapy; a FCBP is a sexually mature woman who: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure
* Patients with a history of prior malignancy are eligible provided there is no active malignancy and a low expectation of recurrence within 6 months

Exclusion Criteria:

* No prior systemic therapy with the exception of bisphosphonates for multiple myeloma
* Prior glucocorticosteroid therapy for the treatment of multiple myeloma is not permitted; prior systemic glucocorticosteroid use for the treatment of non-malignant disorders is permitted; concurrent use after registration on the study should be restricted to the equivalent of prednisone 10 mg per day; prior or concurrent topical or localized glucocorticosteroid therapy to treat non-malignant comorbid disorders is permitted
* Patients must not have active, uncontrolled seizure disorder; patients must have had no seizures in the last 6 months
* Patients must not have uncontrolled intercurrent illness including uncontrolled hypertension, symptomatic congestive heart failure, unstable angina, uncontrolled cardiac arrhythmia, uncontrolled psychiatric illness or social situation that would limit compliance with the study, or a prior history of Stevens Johnson syndrome
* Patients with smoldering myeloma or monoclonal gammopathy of undetermined significance are not eligible
* Patients must not have grade 2 or higher peripheral neuropathy due to other medical conditions at the time of randomization
* Patients must not have active, uncontrolled infection
* Patients must not have a history of current or previous deep vein thrombosis or pulmonary embolism regardless of whether or not the patient is receiving anticoagulation therapy

  * For patients registered prior to activation of Addendum # 6; patients must be willing and able to take prophylaxis with either aspirin at 325 mg/day or alternative prophylaxis with either low molecular weight heparin or Coumadin
  * For patients registered after activation of Addendum # 6; patients entering the expansion phase of the protocol, which tests anticoagulant prophylaxis, must be able and willing to be randomized between aspirin at 325 mg/day and Coumadin
* Female patients MUST NOT be pregnant or breastfeeding; due to the potential teratogenic properties of CC 5013, and the known teratogenicity associated with thalidomide, the use of these drugs in this patient population is ABSOLUTELY CONTRAINDICATED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2004-11-03 (Actual); Primary Completion 2008-11-30 (Actual); Study Completion 2026-10-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: S. V Rajkumar, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (138):
- United States (138):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Saint Jude Medical Center, Fullerton, California
  - El Camino Hospital, Mountain View, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Martin Hospital South, Stuart, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - HealthAlliance Hospital - Leominster, Leominster, Massachusetts
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Union Square, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Mission Hospital, Asheville, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Kaiser Permanente Northwest, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple Health - Chestnut Hill Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - McLeod Regional Medical Center, Florence, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Medical Center-First Hill, Seattle, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin

REFERENCES:
- [Derived] Baker A, Braggio E, Jacobus S, Jung S, Larson D, Therneau T, Dispenzieri A, Van Wier SA, Ahmann G, Levy J, Perkins L, Kim S, Henderson K, Vesole D, Rajkumar SV, Jelinek DF, Carpten J, Fonseca R. Uncovering the biology of multiple myeloma among African Americans: a comprehensive genomics approach. Blood. 2013 Apr 18;121(16):3147-52. doi: 10.1182/blood-2012-07-443606. Epub 2013 Feb 19. PMID 23422747
- [Derived] Kumar SK, Uno H, Jacobus SJ, Van Wier SA, Ahmann GJ, Henderson KJ, Callander NS, Haug JL, Siegel DS, Greipp PR, Fonseca R, Rajkumar SV. Impact of gene expression profiling-based risk stratification in patients with myeloma receiving initial therapy with lenalidomide and dexamethasone. Blood. 2011 Oct 20;118(16):4359-62. doi: 10.1182/blood-2011-03-342089. Epub 2011 Aug 22. PMID 21860025
- [Derived] Rajkumar SV, Jacobus S, Callander NS, Fonseca R, Vesole DH, Williams ME, Abonour R, Siegel DS, Katz M, Greipp PR; Eastern Cooperative Oncology Group. Lenalidomide plus high-dose dexamethasone versus lenalidomide plus low-dose dexamethasone as initial therapy for newly diagnosed multiple myeloma: an open-label randomised controlled trial. Lancet Oncol. 2010 Jan;11(1):29-37. doi: 10.1016/S1470-2045(09)70284-0. Epub 2009 Oct 21. PMID 19853510

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened on October 26, 2004 and was closed on June 1, 2007 with a total accrual of 452 patients enrolled from 6 groups and 77 institutions.
Groups:
- Arm I (Lenalidomide, Dexamethasone): Patients receive oral lenalidomide once daily on days 1-21, oral aspirin (or other deep vein thrombosis prophylaxis at the discretion of the principal investigator) once daily on days 1-28, and standard-dose oral dexamethasone once daily on days 1-4, 9-12, and 17-20. Patients with minimal response or no response after 4 cycles of treatment could register for Step 2 treatment with thalidomide and high-dose dexamethasone. Thalidomide was given orally once daily on days 1-28, and dexamethasone once daily on days 1-4, 9-12, and 17-20 for 4 cycles.
- Arm II (Lenalidomide, Low-dose Dexamethasone): Patients receive oral lenalidomide and acetylsalicylic acid as in arm I and low-dose oral dexamethasone once daily on days 1, 8, 15, and 22. Patients with minimal response or no response after 4 cycles of treatment could register for Step 2 treatment with thalidomide and low-dose dexamethasone. Thalidomide was given orally once daily on days 1-28, and dexamethasone once daily on days 1, 8, 15, and 22 for 4 cycles.
- Arm III (Expansion; Lenalidomide, Dexamethasone, Aspirin): Patients receive oral lenalidomide once daily on days 1-21, oral aspirin (or other deep vein thrombosis prophylaxis at the discretion of the principal investigator) once daily on days 1-28, and standard-dose oral dexamethasone once daily on days 1-4, 9-12, and 17-20. After 4 cycles of treatment, patients may discontinue treatment or continue until progression.
- Arm IV (Expansion; Lenalidomide, Dexamethasone, Coumadin): Patients receive oral lenalidomide once daily on days 1-21, oral aspirin (or other deep vein thrombosis prophylaxis at the discretion of the principal investigator) once daily on days 1-28, and standard-dose oral dexamethasone once daily on days 1-4, 9-12, and 17-20. After 4 cycles of treatment, patients may discontinue treatment. For patients continuing therapy beyond 4 cycles, coumadin was discontinued and aspirin was given instead.
Period: Step 1
Arm/Group | Arm I (Lenalidomide, Dexamethasone) | Arm II (Lenalidomide, Low-dose Dexamethasone) | Arm III (Expansion; Lenalidomide, Dexamethasone, Aspirin) | Arm IV (Expansion; Lenalidomide, Dexamethasone, Coumadin)
Started | 223 | 222 | 4 | 3
Treated | 223 | 220 | 4 | 3
Eligible | 214 (Some patients were considered eligible at registration but found ineligible in the analysis.) | 208 (Some patients were considered eligible at registration but found ineligible in the analysis.) | 4 | 3
Completed | 52 | 49 | 0 | 0
Not Completed | 171 | 173 | 4 | 3
Not completed — Progressive disease | 33 | 35 | 2 | 1
Not completed — Adverse Event | 56 | 37 | 0 | 1
Not completed — Death | 8 | 5 | 0 | 1
Not completed — Withdrawal by Subject | 14 | 11 | 0 | 0
Not completed — Physician Decision | 5 | 2 | 0 | 0
Not completed — Alternative therapy | 31 | 43 | 1 | 0
Not completed — Other disease | 2 | 1 | 1 | 0
Not completed — Never started treatment | 0 | 2 | 0 | 0
Not completed — Still on treatment as of this analysis | 14 | 27 | 0 | 0
Not completed — Knee surgery | 1 | 0 | 0 | 0
Not completed — Complications | 1 | 0 | 0 | 0
Not completed — Cannot comply due to other tx | 0 | 1 | 0 | 0
Not completed — Both patient and physician's decision | 2 | 1 | 0 | 0
Not completed — Incorrect disease assessment | 2 | 0 | 0 | 0
Not completed — Off treatment for > specified timeframe | 1 | 1 | 0 | 0
Not completed — Declining performance status | 0 | 1 | 0 | 0
Not completed — Insurance issue | 0 | 1 | 0 | 0
Not completed — Rising paraprotein | 0 | 1 | 0 | 0
Not completed — Referred to other physicians | 0 | 1 | 0 | 0
Not completed — Criteria to continue treatment not met | 0 | 1 | 0 | 0
Not completed — Misinterpretation of lab data | 0 | 1 | 0 | 0
Not completed — Patient fell with fracture | 1 | 0 | 0 | 0
Not completed — Not documented | 0 | 1 | 0 | 0
Period: Step 2
Arm/Group | Arm I (Lenalidomide, Dexamethasone) | Arm II (Lenalidomide, Low-dose Dexamethasone) | Arm III (Expansion; Lenalidomide, Dexamethasone, Aspirin) | Arm IV (Expansion; Lenalidomide, Dexamethasone, Coumadin)
Started | 5 (Step 2 treatment was an option but not required for patients who ended step 1 treatment.) | 15 (Step 2 treatment was an option but not required for patients who ended step 1 treatment.) | 0 | 0
Treated | 4 | 14 | 0 | 0
Eligible | 2 (Some patients were considered eligible at registration but found ineligible in the analysis.) | 9 (Some patients were considered eligible at registration but found ineligible in the analysis.) | 0 | 0
Completed | 0 | 5 | 0 | 0
Not Completed | 5 | 10 | 0 | 0
Not completed — Disease progression | 1 | 4 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Alternative therapy | 1 | 2 | 0 | 0
Not completed — Never started treatment | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Lenalidomide, Dexamethasone): Patients receive oral lenalidomide once daily on days 1-21, oral aspirin (or other deep vein thrombosis prophylaxis at the discretion of the principal investigator) once daily on days 1-28, and standard-dose oral dexamethasone once daily on days 1-4, 9-12, and 17-20. Patients with minimal response or no response after 4 cycles of treatment could register for Step 2 treatment with thalidomide and high-dose dexamethasone. Thalidomide was given orally once daily on days 1-28, and dexamethasone once daily on days 1-4, 9-12, and 17-20 for 4 cycles.
  As the expansion phase was a substudy terminated early with only 7 patients enrolled, the clinical results presented are mainly for the first phase only. Toxicity data are available for both the first phase and the expansion phase.
- Arm II (Lenalidomide, Low-dose Dexamethasone): Patients receive oral lenalidomide and acetylsalicylic acid as in arm I and low-dose oral dexamethasone once daily on days 1, 8, 15, and 22. Patients with minimal response or no response after 4 cycles of treatment could register for Step 2 treatment with thalidomide and low-dose dexamethasone. Thalidomide was given orally once daily on days 1-28, and dexamethasone once daily on days 1, 8, 15, and 22 for 4 cycles.
  As the expansion phase was a substudy terminated early with only 7 patients enrolled, the clinical results presented are mainly for the first phase only. Toxicity data are available for both the first phase and the expansion phase.
- Total: Total of all reporting groups
Arm/Group | Arm I (Lenalidomide, Dexamethasone) | Arm II (Lenalidomide, Low-dose Dexamethasone) | Total
Number analyzed (Participants) | 223 | 222 | 445
Age, Continuous [Median (Full Range); unit: years] | 66 [36 to 87] | 65 [35 to 85] | 65 [35 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 101 | 192
  Male | 132 | 121 | 253

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Objective Response (First Phase, Step 1)
Description: Objective response is defined as either complete response (CR) or partial response (PR). Patients who have complete disappearance of an M-protein and no evidence of myeloma in the bone marrow are considered to have CR. PR requires all the following: (1) ≥50% reduction in the level of the serum monoclonal paraprotein. (2) Reduction in 24-hour urinary light chain excretion either by ≥90% or to <200 mg. (3)For patients with non-secretory (or oligosecretory) myeloma only, a ≥50% reduction in plasma cells in a bone marrow aspirate and on trephine biopsy must be documented. (4)50% reduction in size of soft tissue plasmacytoma (by radiography or clinical examination). (5) No increase in the number or size of lytic bone lesions (development of a compression fracture does not exclude response).
  As the expansion phase was a substudy terminated early with only 7 patients enrolled, the clinical results presented are mainly for the first phase only.
Time Frame: Assessed every 4 weeks for 16 weeks during Step 1
Population: Only eligible patients were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm I (Lenalidomide, Dexamethasone) | Arm II (Lenalidomide, Low-dose Dexamethasone)
Number analyzed (Participants) | 214 | 208
Proportion of patients | 0.79 [0.729 to 0.842] | 0.683 [0.615 to 0.745]
Statistical Analysis 1: Comparison: Arm I (Lenalidomide, Dexamethasone) vs Arm II (Lenalidomide, Low-dose Dexamethasone); The study was designed to determine if a reduced dose of dexamethasone in combination with CC-5013 reduced toxicity rate without reducing response rate. The standard-dose response was expected to be 70%. The low dose would be deemed unacceptable if the difference in response rate between arms was >=15%. The null hypothesis was that response rates were equal and the alternative was that the low-dose response was no worse than 55%. The design had a 1-sided 0.10 type I error rate and 95% power; Test type: Non-Inferiority or Equivalence — The low-dose response would be considered unacceptable if the difference in response rates was 15% or greater (the upper confidence limit exceeds the 15% acceptable difference) regardless of a decrease in toxicity rate; Difference in response rate between arms = 0.107, 80% CI 2-sided [0.052 to 0.162]

2. Secondary Outcome: Proportion of Patients With Objective Response (First Phase, Step 2)
Description: as for outcome 1
Time Frame: Assessed every 4 weeks for 16 weeks during Step 2
Population: Only eligible patients were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm I (Lenalidomide, Dexamethasone) | Arm II (Lenalidomide, Low-dose Dexamethasone)
Number analyzed (Participants) | 2 | 9
Proportion of patients | 0 [0.0 to 0.842] | 0 [0.0 to 0.336]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment.
Groups:
- Arm I (Lenalidomide, Dexamethasone) Step 1: Patients receive oral lenalidomide once daily on days 1-21, oral aspirin (or other deep vein thrombosis prophylaxis at the discretion of the principal investigator) once daily on days 1-28, and standard-dose oral dexamethasone once daily on days 1-4, 9-12, and 17-20. Patients with minimal response or no response after 4 cycles of treatment could register for Step 2 treatment with thalidomide and high-dose dexamethasone. Thalidomide was given orally once daily on days 1-28, and dexamethasone once daily on days 1-4, 9-12, and 17-20 for 4 cycles.
- Arm II (Lenalidomide, Low-dose Dexamethasone) Step 1: Patients receive oral lenalidomide and acetylsalicylic acid as in arm I and low-dose oral dexamethasone once daily on days 1, 8, 15, and 22. Patients with minimal response or no response after 4 cycles of treatment could register for Step 2 treatment with thalidomide and low-dose dexamethasone. Thalidomide was given orally once daily on days 1-28, and dexamethasone once daily on days 1, 8, 15, and 22 for 4 cycles.
- Arm I (Lenalidomide, Dexamethasone) Step 2: Arm I patients with minimal response or no response after 4 cycles of treatment in Step 1 could register for Step 2 treatment with thalidomide and high-dose dexamethasone. Thalidomide was given orally once daily on days 1-28, and dexamethasone once daily on days 1-4, 9-12, and 17-20 for 4 cycles.
- Arm II (Lenalidomide, Low-dose Dexamethasone) Step 2: Arm II patients with minimal response or no response after 4 cycles of treatment in Step 1 could register for Step 2 treatment with thalidomide and low-dose dexamethasone. Thalidomide was given orally once daily on days 1-28, and dexamethasone once daily on days 1, 8, 15, and 22 for 4 cycles.
Arm/Group | Arm I (Lenalidomide, Dexamethasone) Step 1 | Arm II (Lenalidomide, Low-dose Dexamethasone) Step 1 | Arm I (Lenalidomide, Dexamethasone) Step 2 | Arm II (Lenalidomide, Low-dose Dexamethasone) Step 2 | Arm III (Expansion; Lenalidomide, Dexamethasone, Aspirin) | Arm IV (Expansion; Lenalidomide, Dexamethasone, Coumadin)
Serious Adverse Events (participants affected / at risk) | 146/223 | 112/220 | 1/4 | 3/14 | 2/4 | 1/3
Other Adverse Events (participants affected / at risk) | 222/223 | 216/220 | 4/4 | 14/14 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Lenalidomide, Dexamethasone) Step 1 (N=223) | Arm II (Lenalidomide, Low-dose Dexamethasone) Step 1 (N=220) | Arm I (Lenalidomide, Dexamethasone) Step 2 (N=4) | Arm II (Lenalidomide, Low-dose Dexamethasone) Step 2 (N=14) | Arm III (Expansion; Lenalidomide, Dexamethasone, Aspirin) (N=4) | Arm IV (Expansion; Lenalidomide, Dexamethasone, Coumadin) (N=3)
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac-ischemia (Cardiac disorders) | 7 | 1 | 0 | 0 | 0 | 0
Cardiac troponin T (cTnT) (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 4 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 2 | 0 | 0 | 0 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 33 | 21 | 0 | 0 | 1 | 1
Fever w/o neutropenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 2 | 0 | 0 | 0 | 0
Rigors/chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 | 9 | 0 | 0 | 0 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Death - sudden death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic glucose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Endocrine-other (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 9 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 2 | 0 | 0 | 0 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4 | 3 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Fistula, Ileum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 0 | 0
Perforation, colon (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Ulcer, gastric (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0 | 1
Gastrointestinal (GI) - other (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Duodenum, hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectum, hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Lung, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hemorrhage-other (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Infection w/ grade 3-4 neutropenia, colon (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infection with grade 3-4 neutropenia, lung (Infections and infestations) | 1 | 4 | 0 | 0 | 0 | 1
Infection with grade 3-4 neutropenia, upper airway (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Infection with grade 3-4 neutropenia, urinary tract (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Infection with grade 0-2 neutropenia, brain (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infection with grade 0-2 neutropenia, bronchus (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Infection with grade 0-2 neutropenia, colon (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infection with grade 0-2 neutropenia, esophagus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infection with grade 0-2 neutropenia, lip/perioral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infection with grade 0-2 neutropenia, lung (Infections and infestations) | 11 | 1 | 0 | 0 | 0 | 0
Infection with grade 0-2 neutropenia, middle ear (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infection with grade 0-2 neutropenia, skin (Infections and infestations) | 6 | 4 | 0 | 0 | 0 | 0
Infection with grade 0-2 neutropenia, urinary tract (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Colon infection with unknown absolute neutrophil count (ANC) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung infection with unknown absolute neutrophil count (ANC) (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0
Wound infection with unknown absolute neutrophil count (ANC) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Opportunistic infection associated with >= Grade 1 lymphopenia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infection with grade 3-4 neutropenia, blood (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0
Infection with grade 0-2 neutropenia, blood (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0
Infection w/ unk ANC blood (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infection - other (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Edema head and neck (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Edema limb (General disorders) | 14 | 3 | 0 | 1 | 1 | 0
Edema trunk/genital (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase (ALT) increased (Investigations) | 6 | 4 | 0 | 0 | 0 | 0
Aspartate aminotransferase (AST) increased (Investigations) | 3 | 2 | 0 | 0 | 0 | 0
Bilirubin increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 16 | 8 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 6 | 4 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 25 | 13 | 0 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 17 | 8 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 12 | 3 | 0 | 0 | 0 | 0
Metabolic/Laboratory - other (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Nonneuropathic extraocular muscle weak (Eye disorders) | 11 | 4 | 0 | 0 | 0 | 0
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 13 | 4 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Central nervous system (CNS) cerebrovascular ischemia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 4 | 2 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 6 | 3 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Extrapyramidal movement (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 7 | 4 | 0 | 0 | 0 | 0
Neuropathy cranial nerves (CN) II vision (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy-motor (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 2 | 3 | 0 | 0 | 0 | 0
Psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Speech impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 4 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 2 | 4 | 0 | 0 | 0 | 0
Vision-blurred (Eye disorders) | 3 | 0 | 0 | 0 | 0 | 0
Abdomen, pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac/heart, pain (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest/thoracic pain NOS (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0
Muscle pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Neuropathic, pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain - other (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 4 | 0 | 0 | 2 | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0 | 0 | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 0 | 0 | 0 | 0
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 4 | 1 | 0 | 0 | 0 | 1
Urinary electrolyte wasting (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 56 | 28 | 0 | 0 | 1 | 0
Vascular-Other (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Lenalidomide, Dexamethasone) Step 1 (N=223) | Arm II (Lenalidomide, Low-dose Dexamethasone) Step 1 (N=220) | Arm I (Lenalidomide, Dexamethasone) Step 2 (N=4) | Arm II (Lenalidomide, Low-dose Dexamethasone) Step 2 (N=14) | Arm III (Expansion; Lenalidomide, Dexamethasone, Aspirin) (N=4) | Arm IV (Expansion; Lenalidomide, Dexamethasone, Coumadin) (N=3)
Fatigue (General disorders) | 132 | 136 | 2 | 10 | 3 | 1
Fever w/o neutropenia (General disorders) | 23 | 12 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 76 | 84 | 0 | 2 | 2 | 1
Sweating (Skin and subcutaneous tissue disorders) | 21 | 18 | 0 | 0 | 0 | 1
Weight gain (Investigations) | 30 | 17 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 18 | 13 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 3 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 8 | 13 | 0 | 0 | 0 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 15 | 32 | 0 | 0 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 36 | 60 | 0 | 1 | 1 | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 28 | 18 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 74 | 87 | 3 | 8 | 0 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 36 | 45 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 23 | 19 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 49 | 45 | 0 | 1 | 1 | 2
Taste disturbance (Nervous system disorders) | 20 | 17 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 13 | 13 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0
Infection with grade 0-2 neutropenia, bladder (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Opportunistic infection associated with >= Grade 1 lymphopenia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Edema, limb (General disorders) | 90 | 69 | 2 | 4 | 1 | 1
Alkaline phosphatase increased (Investigations) | 56 | 50 | 0 | 2 | 0 | 0
ALT increased (Investigations) | 78 | 67 | 0 | 0 | 2 | 0
AST increased (Investigations) | 50 | 51 | 1 | 1 | 3 | 0
Bilirubin increased (Investigations) | 24 | 24 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 13 | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 130 | 114 | 0 | 3 | 3 | 2
Creatinine increased (Investigations) | 57 | 58 | 0 | 2 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 153 | 151 | 2 | 7 | 2 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 18 | 10 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 17 | 16 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 68 | 67 | 0 | 1 | 1 | 2
Hypernatremia (Metabolism and nutrition disorders) | 13 | 22 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 76 | 59 | 0 | 1 | 2 | 1
Nonneuropathic extraocular muscle weak (Eye disorders) | 51 | 27 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 45 | 25 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 19 | 5 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 54 | 42 | 0 | 0 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 83 | 68 | 1 | 4 | 0 | 0
Tremor (Nervous system disorders) | 45 | 37 | 2 | 2 | 0 | 0
Vision - blurred (Eye disorders) | 39 | 36 | 0 | 0 | 0 | 1
Abdomen, pain (General disorders) | 10 | 6 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 22 | 1 | 0 | 1 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 13 | 11 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 21 | 18 | 0 | 0 | 0 | 0
Muscle pain (Musculoskeletal and connective tissue disorders) | 14 | 18 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 40 | 38 | 1 | 2 | 0 | 0
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 6 | 3 | 0 | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 7 | 0 | 1 | 0 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 9 | 8 | 0 | 1 | 0 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 7 | 9 | 0 | 1 | 0 | 0
Ulcer, gastric (Gastrointestinal disorders) | 5 | 8 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 4 | 1 | 0 | 2 | 0 | 0
Confusion (Psychiatric disorders) | 11 | 8 | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 5 | 7 | 0 | 3 | 0 | 0
Pain NOS (General disorders) | 0 | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less